CLINICAL TRIAL: NCT04572087
Title: Ameliorating Cognitive Control in Binge Eating Disorder by Electrical Brain Stimulation
Brief Title: Ameliorating Cognitive Control in Binge Eating Disorder
Acronym: ACCElect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Katrin Giel (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Katrin Giel, Prof. Dr., University Hospital Tuebingen
Organization: University Hospital Tuebingen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GI 878/4-1; PL 525/7-1 (Other Grant/Funding Number: Deutsche Forschungsgemeinschaft)
Record Dates: First submitted 2020-09-16; First posted 2020-10-01 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2021-09

CONDITIONS: Binge-Eating Disorder
Keywords: Brain stimulation; cognitive control; behavioral training; binge eating disorder; response inhibition; eye tracking; eating disorder; impulsivity
MeSH Terms: conditions — Binge-Eating Disorder; Feeding and Eating Disorders; Impulsive Behavior

STUDY DESIGN:
Intervention Model Description: After the baseline measure (T0) without tDCS, participants are randomized to either the group that receives 6 training sessions (T1-T6) with 2 milliampere (ma) anodal tDCS to the right dlPFC or the group that receives 6 training sessions and sham tDCS.
  After the six training sessions within 2 weeks a post measurement concerning task performance (T7) without tDCS takes place. 4 Weeks after treatment, the diagnostic post measurement (T8) will be executed. 3 months later, a follow-up via phone (T9) will be done.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants as well as the experimenters are blinded to the treatment group by using a unique 5-digit code for each participant which activates either verum or sham stimulation. The participants and experimenters are blinded to the randomisation condition as current in the sham condition is applied for 40 seconds at the beginning of each training session and during this time, no training of the cognitive control task is done. As participants perceive typical sensations of tDCS (e.g. tingling) and tDCS electrodes are actually mounted, this is considered as a valid placebo control.
  The PIs and the biostatistician from the external ICEAB who is doing the statistical analysis are blinded as well until the end of the analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Control Training + Verum stimulation (Experimental): This arm consists of the cognitive control training (six sessions) combined with 2mA anodal tDCS over the right dlPFC (F4) during the training for 20 minutes.
  Interventions: Other: Behavioral training and verum stimulation
- Cognitive Control Training + Sham stimulation (Active Comparator): This arm consists of cognitive control training (six sessions) with sham-tDCS. 2 mA Sham-tDCS (40 seconds of tDCS) is applied to the right dlPFC (F4) before the trainings starts.
  Interventions: Other: Behavioral training and sham stimulation

INTERVENTIONS:
Other: Behavioral training and verum stimulation — Cognitive control training and verum tDCS
  Arms: Cognitive Control Training + Verum stimulation
Other: Behavioral training and sham stimulation — Cognitive control training and sham tDCS
  Arms: Cognitive Control Training + Sham stimulation

SUMMARY:
There is evidence that impairment of impulse regulation is involved in the development and maintenance of eating disorders, especially in Binge Eating Disorder (BED). BED is characterized by recurrent episodes of binge eating with experienced loss of control over eating. Controlling impulsive behaviour, cognitive flexibility, planning and decision making are key abilities of impulse regulation. Some of these impaired cognitive functions are linked to decreased activity of certain brain regions. Transcranial direct current stimulation (tDCS) is a well-established method to alter brain activity. In the current project, we explore if a computer-assisted training programme for patients with BED that is combined with tDCS is feasible and able to ameliorate impulse regulation and impulsive eating behaviour. We hypothesize that the cognitive training programme with additional tDCS will result in a greater decrease of BED symptoms and a stronger increase in impulse regulation skills compared with the cognitive training programme without tDCS by using a placebo stimulation.

DETAILED DESCRIPTION:
Patients with BED form a subgroup of obese patients with a disinhibited eating pattern that is associated with major impairments in cognitive control. The dorsolateral prefrontal cortex (dlPFC) has been identified as a brain region closely tied to cognitive control processes and crucially involved in the control of eating behaviour. This suggests the dlPFC as a target for the modulation of cognitive control processes over eating in BED. This modulation can be achieved by both, a cognitive training task and by noninvasive brain stimulation using tDCS. In studies with healthy normal-weight participants, (1) different cognitive training task enhance control over eating behaviour, (2) tDCS is an effective tool to ameliorate cognitive control processes, and (3) has beneficial effects on motivational aspects of eating behaviour, i.e. food craving. Based on this evidence, we will use a combination of a cognitive control task and tDCS to enhance cognitive control over eating in patients with BED. This is to the best of our knowledge one of the first studies to use tDCS as an intervention to enhance cognitive control over eating in patients with BED.

o Sample size: We will allocate 40 patients in the trial, i.e. 20 patients in each study arm.

o Recruitment: Patients are recruited by announcements, mails to the distributor list of the university hospital, existing databases of patients, and current patients of the university hospital. Patients are screened by a standardized checklist. In- and exclusion criteria are checked during the screening procedure and during the baseline diagnostic before randomisation.

o Standard Operating Procedures: For the recruitment, diagnostic and experimental sessions, Standard Operating Procedures are documented for the experimenter. This includes the order of clinical interviews, questionnaires and operating with the technical measurement instruments. The experimenters are regularly supervised. All adverse events will be listed and severe adverse events will be reported immediately to the PIs.

o Quality assurance plan: Randomized allocation to the stimulation condition (verum vs. sahm) and statistical analyses is done externally by the Institute of Clinical Epidemiology and Applied Biometry, University Tübingen, Germany (ICEAB). Objective technical measurement instruments are mostly used to record data.

o Data checks: Data is recorded mostly by objective technical measurement instruments, so no external monitoring is needed. We will spot check entered questionnaire data, in particular binge eating frequency in the past four weeks will be double checked as this is the primary outcome (PO).

o Source data verification: Data are spot checked by comparing the entries in the source data with the entries in the database. Each PO entry will be double checked. There are pre-defined criteria for entering data into the database.

* Data dictionary:

A data dictionary that contains detailed descriptions of each variable and how to be entered is available.

o Plan for missing data: Missing data and invalid data as well as the reasons will be recorded.

o Statistical analysis plan: A mixed model approach will be used to analyze the PO and secondary outcomes (SOs).

ELIGIBILITY:
Inclusion Criteria:

* BED according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5)
* Legal age
* BMI above 20 kg/m2

Exclusion Criteria:

* Insufficient knowledge of German language
* Current pregnancy or lactation period
* Current or lifetime psychotic disorder, bipolar-I disorder, current substance dependence, suicidality
* Past bariatric surgery
* Severe physical disease which influence weight or eating behaviour (e.g. severe diabetes) or neurologic disease
* Non-removable metal parts in the area of the head
* Pacemaker
* Neuroleptics and benzodiazepine
* impaired vision, ametropia, eye diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
Binge eating frequency | assessed at baseline (T0) and at diagnostic post assessment four weeks after treatment (T8)
  Change of the frequency of Binge eating episodes in the last 4 weeks according to the Eating Disorder Examination Interview (EDE) between baseline (T0) and diagnostic post assessment (T8). The EDE is a validated semi-structured clinical interview.

SECONDARY OUTCOMES:
Binge eating frequency follow-up | assessed at baseline (T0) and at 3 months follow-up (T9)
  Change of the frequency of Binge eating episodes in the last 4 weeks according to EDE between baseline (T0) and 3 months follow up (T9)
antisaccade task | assessed at baseline (T0), the six training sessions within two weeks (T1-T6) and the post measurement of task performance within one week after the training (T7)
  antisaccade task error rate and latency assessed by eye tracking
Go/No-Go task | at baseline (T0) and at the post measurement of task performance within one week after the training (T7)
  Go/No-Go task task error rate and latency
stimulus rating | at baseline (T0) and and the post measurement of task performance within one week after the training (T7)
  one self-developed questionnaire including visual analogue scales (0-10 cm) concerning valence, appetite, wanting, liking of the presented stimuli
Eating disorder pathology (EDE) | assessed at baseline (T0), at diagnostic post assessment four weeks after treatment (T8) and 3 months follow-up (T9)
  assessed by the Eating Disorder Examination (EDE), Range 0-6 with higer scores indication higer eating disorder pathology
eating behaviour (TFEQ) | at baseline (T0), at the post measurement of task performance within one week after the training (T7) and at diagnostic post assessment four weeks after treatment (T8)
  assessed by the Three-factor Eating Questionnaire (TFEQ), Range 0-1 with higher scores indicating more pathological eating behaviour
food craving (FCQ-S) | at baseline (T0), the six training sessions within two weeks (T1-T6) and the post measurement of task performance within one week after the training (T7)
  assessed by the Food Craving Questionnaire, State Version (FCQ-S), Range 1-5 with higher scores indicating higher food craving
impulsive behaviours per week | at baseline (T0), the six training sessions within two weeks (T1-T6), the post measurement of task performance within one week after the training (T7) and at diagnostic post assessment four weeks after treatment (T8)
  assessed by a self-developed process analysis questionnaire, values > 0 (unlimited frequency) with higher scores indicating more impulsive behaviours per week
impulsivity (UPPS) | at baseline (T0) and at diagnostic post assessment four weeks after treatment (T8)
  assessed by the "UPPS Impulsive Behavior Scale" (UPPS), Range 1-4 with higher scores indicating higher impulsivity
well-being (WHO-5) | at baseline (T0), the post measurement of task performance within one week after the training (T7) and at diagnostic post assessment four weeks after treatment (T8)
  assessed by the "WHO (Five) - Well-being Questionnaire" (WHO-5), Range 0-5 with higher scores indicating higher well-being
depressive symptoms (BDI II) | at baseline (T0) and at diagnostic post assessment four weeks after treatment (T8)
  assessed by the Becks Depression Inventory, Version 2 (BDI II), Range 0-3 with higher scores indicating higher depressive symptoms
Body Mass Index (BMI) | at baseline (T0) and at diagnostic post assessment four weeks after treatment (T8)
  computed by objectively assessed weight and height
acceptance and feasibility | from baseline (T0) throughout all measurement points until 3 months follow-up (T9)
  drop-out rate throughout T0 to T9, percentage of included patients from the eligible patients at T0
evaluation of the training programme | assessed at the post measurement of task performance within one week after the training (T7)
  self-developed questionnaire at T7 (Range 1-5 with higher cores indicating more satisfaction with the training programme)

CONTACTS AND LOCATIONS:
Overall Officials: Katrin E Giel, Prof. Dr., Principal Investigator — University Hospital Tübingen; Christian Plewnia, Prof. Dr., Principal Investigator — University Hospital Tübingen
Locations (1):
- University Hospital Tübingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Max SM, Plewnia C, Zipfel S, Giel KE, Schag K. Combined antisaccade task and transcranial direct current stimulation to increase response inhibition in binge eating disorder. Eur Arch Psychiatry Clin Neurosci. 2021 Feb;271(1):17-28. doi: 10.1007/s00406-020-01164-5. Epub 2020 Jul 13. PMID 32661703
- [Background] Schag K, Ince B, Zipfel S, Max S, Plewnia C, Giel K. [Non-Invasive Brain Stimulation in the Treatment of Eating Disorders - A Narrative Review]. Psychother Psychosom Med Psychol. 2020 Jun;70(6):246-251. doi: 10.1055/a-1156-8899. Epub 2020 Jun 9. German. PMID 32516813
- [Background] Giel KE, Schag K, Martus P, Max SM, Plewnia C. Ameliorating cognitive control in patients with binge eating disorder by electrical brain stimulation: study protocol of the randomized controlled ACCElect pilot trial. J Eat Disord. 2022 Feb 19;10(1):26. doi: 10.1186/s40337-022-00544-7. PMID 35183261
- See also: research information of the University Tübingen, Germany — https://fit.uni-tuebingen.de/Project/Details?id=5389